CLINICAL TRIAL: NCT03763838
Title: Acupressure for Fatigue in Ovarian Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: UMCC 2018.130; HUM00143509 (Other: University of Michigan); W81XWH1810180 (Other Grant/Funding Number: Defense, Department of-Army, Department of the)
Record Dates: First submitted 2018-12-03; First posted 2018-12-04 (Actual); Results first posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Fatigue; Ovarian Cancer
Keywords: Acupressure
MeSH Terms: conditions — Fatigue; Ovarian Neoplasms | interventions — Acupressure; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants in the "standard of care" arm will not be blinded; however, the two self-acupressure arms will be blinded as to which acupressure treatment they have been randomized. All study staff and researchers will remain blinded until after the completion of data analyses.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupressure plus standard of care (Experimental): Using AcuWand, participants will apply acupressure to points that are known to affect physiology. Participants will also receive standard of care.
  Interventions: Other: Acupressure; Other: Standard of Care
- Sham acupressure plus standard of care (Sham Comparator): Using AcuWand, participants will apply acupressure to points that are not known to affect physiology. Participants will also receive standard of care.
  Interventions: Other: Sham acupressure; Other: Standard of Care
- Standard of care (Other): Participants will receive standard of care only.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Acupressure — Six weeks of daily self-administered relaxing acupressure. Instructions will be provided for how to perform acupressure on self. A tool (AcuWand) will be provided to help participants apply the right amount of pressure on the appropriate points on their bodies. These are points that are recognized as effective in Traditional Chinese Medicine (TCM).
  Arms: Acupressure plus standard of care
Other: Sham acupressure — Six weeks of daily self-administered sham acupressure. Instructions will be provided for how to perform acupressure on self. A tool (AcuWand) will be provided to help participants apply the right amount of pressure; however, the points that participants are instructed to use are not known to have any effect on the body.
  Arms: Sham acupressure plus standard of care
Other: Standard of Care — Fatigue management provided by participants' health care providers.

SUMMARY:
The purpose of this study is to see if accupressure can help reduce the severity of fatigue experienced by ovarian cancer patients. Acupressure involves applying mild to moderate physical pressure by fingers, hand or a device to specific points on the skin to try to bring about a change in the body's functioning, in this case relief from chronic fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 21 and older
* Diagnosis of ovarian cancer, stages I to IV
* Have average persistent fatigue defined a >=4 on the Brief Fatigue Inventory.
* Fatigue must have started at or after the diagnosis of ovarian cancer
* Completed all primary cancer treatments (surgery, chemotherapy at least 6 months prior), except maintenance therapies
* No other planned interventions for fatigue other than current stable medication

Exclusion Criteria:

* Medically unstable
* Acupuncture or acupressure receipt in past year
* Have a diagnosis of untreated mood disorder, e.g., bipolar or major depressive disorder
* Have a current diagnosis of anemia
* Have a current untreated diagnosis of hypothyroidism
* Have an initiation, a cessation or change of treatment of any chronic medications, dietary supplements, behavioral therapy, physical therapy, etc., or any planned change of medications, supplements or therapies during the study
* Have the possibility of becoming pregnant

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanna M Zick, ND, MPH, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zick SM, Chen D, Harris RE, Kruger G, Runyon A, Sen A, Snyder S, Pearce CL. Self-Acupressure for Fatigue in Patients Surviving Ovarian Cancer: A Randomized Clinical Trial. JAMA Netw Open. 2026 Feb 2;9(2):e2556357. doi: 10.1001/jamanetworkopen.2025.56357. PMID 41642626
- [Derived] Zick SM, Kruger G, Harte S, Sen A, Harris RE, Pearce CL. Acupressure for Cancer-fatigue in Ovarian Cancer Survivor (AcuOva) Study: A community-based clinical trial study protocol examining the impact of self-acupressure on persistent cancer-related fatigue in ovarian cancer survivors. Contemp Clin Trials. 2021 Aug;107:106477. doi: 10.1016/j.cct.2021.106477. Epub 2021 Jun 10. PMID 34119716

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Acupressure plus standard of care- 58 participants allocated, 5 participants did not start treatment.
  Sham plus standard of care- 58 participants allocated, 2 participants did not start treatment.
  Standard of care- 55 participants allocated, 4 participants did not start treatment.
Period: Overall Study
Arm/Group | Acupressure Plus Standard of Care | Sham Acupressure Plus Standard of Care | Standard of Care
Started | 58 | 58 | 55
Completed | 37 | 40 | 46
Not Completed | 21 | 18 | 9
Not completed — Lost to Follow-up | 12 | 9 | 5
Not completed — Withdrawal by Subject | 4 | 3 | 0
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Disease Reoccurrence | 0 | 2 | 0
Not completed — participants did not start treatment. | 5 | 2 | 4

BASELINE CHARACTERISTICS:
Population: Including all subjects who were randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Acupressure Plus Standard of Care | Sham Acupressure Plus Standard of Care | Standard of Care | Total
Number analyzed (Participants) | 58 | 58 | 55 | 171
Age, Customized [Mean (Standard Deviation); unit: years] | 57 (10) | 55 (12) | 57 (12) | 57 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 58 | 55 | 171
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 2
  Black or African American | 2 | 1 | 1 | 4
  White | 51 | 51 | 45 | 147
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 3 | 5 | 5 | 13
Region of Enrollment [Number; unit: participants]
  United States | 58 | 58 | 55 | 171

OUTCOME MEASURES:

1. Primary Outcome: Change in Level of Fatigue at Week 6
Description: Self-reported on the Brief Fatigue Inventory (BFI). The Brief Fatigue Inventory (BFI) uses a scale of 0 to 10 for each item, with 0 representing "no fatigue" and 10 representing "fatigue as bad as you can imagine". Scores are then categorized as mild (1-3), moderate (4-6), and severe (7-10). The global BFI score is calculated as the average of all items, and a score of 7 or greater is considered clinically significant.
Time Frame: Baseline to week 6
Population: evaluable patients at week 6
Measure: Mean (95% Confidence Interval); unit: mean score
Arm/Group | Acupressure Plus Standard of Care | Sham Acupressure Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 41 | 45 | 51
mean score
  Baseline | 5.57 [5.09 to 6.06] | 5.30 [4.81 to 5.79] | 5.38 [4.91 to 5.85]
  Week 6 | 3.52 [3.02 to 4.01] | 4.06 [3.60 to 4.53] | 4.96 [4.52 to 5.40]

2. Primary Outcome: Change in Level of Fatigue up to Week 24
Description: as for outcome 1
Time Frame: Baseline up to week 24
Population: evaluable patients at 24 weeks
Measure: Mean (95% Confidence Interval); unit: mean score
Arm/Group | Acupressure Plus Standard of Care | Sham Acupressure Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 37 | 40 | 46
mean score
  Baseline | 5.57 [5.09 to 6.06] | 5.30 [4.81 to 5.79] | 5.38 [4.91 to 5.85]
  Week 24 | 3.55 [2.81 to 4.29] | 4.09 [3.36 to 4.82] | 5.15 [4.63 to 5.68]

3. Secondary Outcome: Change in Quality of Life at Week 6
Description: Self-reported on the Functional Assessment of Cancer Therapy Ovarian (FACT-O). The FACT-O is a questionnaire used to assess the quality of life in women with ovarian cancer. It includes 7 items, each scored from 0 to 4, with higher scores representing a more positive quality of life. Mean scores are reported by arm and timepoint. score range of 0-28.
Time Frame: Baseline to week 6
Population: number of patients evaluable at 6 weeks
Measure: Mean (95% Confidence Interval); unit: mean score
Arm/Group | Acupressure Plus Standard of Care | Sham Acupressure Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 53 | 56 | 51
mean score
  Baseline | 9.32 [8.33 to 10.31] | 9.73 [8.77 to 10.70] | 8.59 [7.58 to 9.60]
  Week 6 | 8.26 [7.20 to 9.33] | 9.31 [8.28 to 10.33] | 8.67 [7.65 to 9.69]

4. Secondary Outcome: Change in Quality of Life up to Week 24
Description: as for outcome 3
Time Frame: Baseline up to week 24
Population: Number of evaluable patients at 24 weeks
Measure: Mean (95% Confidence Interval); unit: mean score
Arm/Group | Acupressure Plus Standard of Care | Sham Acupressure Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 37 | 40 | 45
mean score
  Baseline | 9.32 [8.33 to 10.31] | 9.73 [8.77 to 10.70] | 8.59 [7.58 to 9.60]
  Week 24 | 8.06 [6.97 to 9.15] | 8.58 [7.53 to 9.62] | 8.16 [7.12 to 9.19]

5. Secondary Outcome: Change in Sleep Quality at Week 6
Description: Self-reported on the Pittsburgh Sleep Quality Index (PSQI). The Pittsburgh Sleep Quality Index (PSQI) yields a global score ranging from 0 to 21, with higher scores indicating poorer sleep quality.
Time Frame: Baseline to week 6
Population: evaluable patients at 6 weeks
Measure: Mean (95% Confidence Interval); unit: mean score
Arm/Group | Acupressure Plus Standard of Care | Sham Acupressure Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 40 | 45 | 50
mean score
  Baseline | 9.32 [8.33 to 10.31] | 9.73 [8.77 to 10.70] | 8.59 [7.58 to 9.60]
  Week 6 | 8.26 [7.20 to 9.33] | 9.31 [8.28 to 10.33] | 8.67 [7.65 to 9.69]

6. Secondary Outcome: Change in Sleep Quality up to Week 24
Description: as for outcome 5
Time Frame: Baseline up to week 24
Population: evaluable patients at 24 weeks
Measure: Mean (95% Confidence Interval); unit: mean score
Arm/Group | Acupressure Plus Standard of Care | Sham Acupressure Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 37 | 40 | 45
mean score
  Baseline | 9.32 [8.33 to 10.31] | 9.73 [8.77 to 10.70] | 8.59 [7.58 to 9.60]
  Week 24 | 8.06 [6.97 to 9.15] | 8.58 [7.53 to 9.62] | 8.16 [7.12 to 9.19]

ADVERSE EVENTS:
Time Frame: All adverse event data (serious and non-serious) collected from the time of the initial study treatment administration through the follow up visit at week 6.
Arm/Group | Acupressure Plus Standard of Care | Sham Acupressure Plus Standard of Care | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/56 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/53 | 1/56 | 0/51
Other Adverse Events (participants affected / at risk) | 0/53 | 1/56 | 0/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acupressure Plus Standard of Care (N=53) | Sham Acupressure Plus Standard of Care (N=56) | Standard of Care (N=51)
Guillain-Barré syndrome (GBS) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acupressure Plus Standard of Care (N=53) | Sham Acupressure Plus Standard of Care (N=56) | Standard of Care (N=51)
rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-01-23): https://cdn.clinicaltrials.gov/large-docs/38/NCT03763838/Prot_SAP_000.pdf
  • Informed Consent Form (2023-11-13): https://cdn.clinicaltrials.gov/large-docs/38/NCT03763838/ICF_001.pdf